CLINICAL TRIAL: NCT06128616
Title: Efficacy of Extracorporeal Shock Wave Therapy Integrated to Combined Treatment of Botulinum Toxin A and Serial Casting in Children With Cerebral Palsy
Brief Title: Efficacy of Extracorporeal Shock Wave Therapy in Children With Cerebral Palsy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK/16.bI.06
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spasticity/Paresis; Cerebral Palsy
Keywords: Spasticity; Cerebral Palsy; Botulinum toxin A; Extracorporeal Shock Wave Therapy; Casting
MeSH Terms: conditions — Muscle Spasticity; Paresis; Cerebral Palsy | interventions — Botulinum Toxins, Type A; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT Group (Experimental): Patients treated by BoNT-A, intermittent SC and ESWT, whom received either PT or OT
  Interventions: Device: ESWT; Drug: Botulinum Toxin Type A; Other: Serial Casting; Behavioral: Physical Therapy; Behavioral: Occupational Therapy
- Control Group (Active Comparator): Patients treated by BoNT-A, and intermittent SC, whom received either PT or OT
  Interventions: Drug: Botulinum Toxin Type A; Other: Serial Casting; Behavioral: Physical Therapy; Behavioral: Occupational Therapy

INTERVENTIONS:
Device: ESWT — Extracorporeal Shock Wave Therapy
  Arms: ESWT Group
Drug: Botulinum Toxin Type A — Botulinum Toxin Type A
  Other Names: Botox
Other: Serial Casting — Serial Casting
Behavioral: Physical Therapy — Physical Therapy
Behavioral: Occupational Therapy — Occupational Therapy

SUMMARY:
Spastic plantar and palmar flexion deformities are very common in children with cerebral palsy (CP). These deformities usually involve spasticity of the plantar or palmar muscle complexes, weakness of the antagonist dorsiflexor muscles of the ankle or wrist, and also involve soft tissue/muscle contractures and require a multimodal treatment approach. Physical therapy (PT), occupational therapy (OT), serial casting (SC), and botulinum toxin A (BoNT-A) injections had shown positive results in both of these deformities. Recent systematic reviews and meta-analyses showed that extracorporeal shock wave therapy (ESWT) is effective in reducing spasticity, pain intensity, and increasing range of motion and motor function when combined with PT or BoNT-A injections in neurological conditions like stroke, CP, multiple sclerosis. ESWT can be a complimentary therapy to obtain an earlier efficacy, better efficacy, a sustained effect for a longer period, and less adverse events. The objective of this study was to show the effects of ESWT when combined with intermittent SC, BoNT-A injections and PT or OT on spasticity, passive range of motion (pROM) of children with CP having spastic equinus foot deformity or wrist palmar flexion deformity.

DETAILED DESCRIPTION:
Spasticity is one of the most common motor disorder which may slowly cause soft tissue contractures in children with CP. Spastic plantar and palmar flexion deformities are very common in children with CP. These deformities usually involve spasticity of the plantar or palmar muscle complexes, weakness of the antagonist dorsiflexor muscles of the ankle or wrist, and also involve soft tissue/muscle contractures. PT, OT, SC, and BoNT-A injections had shown positive results in both of these deformities. Skin irritation or breakdown, painful episodes, oedema, tendonitis, weakness, stiffness are some of the side effects reported after SC. Moreover casting especially when prolonged might complicate activities of daily living for instance by increasing the risk of falls or causing problems in bathing. Recent evidence from literature favors early, goal oriented, activity based, intensive, repetitive motor trainings in enriched environments to optimize neuroplasticity in children with CP. Prolonged SC might also interfere with these activity based, intensive rehabilitation options for upper extremity. In order to overcome the issues with patient compliance, side effects and combined treatment options an intermittent SC model was developed and used both for children with CP presenting equines foot deformity or palmar flexion deformity. Combined management of intermittent SC, and BoNT-A injections had shown better results compared to either treatment alone in both of these deformities. Recent systematic reviews and meta-analyses showed that ESWT is effective in reducing spasticity, pain intensity, and increasing range of motion and motor function when combined with PT or BoNT-A injections in neurological conditions like stroke, CP, multiple sclerosis. ESWT can be a complementary therapy to obtain an earlier efficacy, better efficacy, a sustained effect for a longer period, and less adverse events.

The objective of this study was to show the effects of ESWT when combined with intermittent SC, BoNT-A injections and PT or OT on spasticity, passive range of motion (pROM) of children with CP having spastic equinus foot deformity or wrist palmar flexion deformity.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of CP according to Rosenbaum criteria, presenting plantar or palmar flexion deformity, having a Modified Ashworth Scale score of 3 in plantar or palmar flexor muscle groups, being scheduled for BoNT-A treatment, intermittent serial casting and physical or occupational therapy

Exclusion Criteria:

* Having cognitive dysfunction, having a history of orthopedic surgery, presenting significant dystonia, having vascular disease, fracture, or dislocation

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline Tardieu XV3 angle | Post-treatment weeks 4-6
  Spasticity measurement
Mean change from baseline passive range of movement | Post-treatment weeks 12-20
  Soft tissue contracture measurement

SECONDARY OUTCOMES:
Goal Attainment Scale-Light | Post-treatment weeks 4-12-20
  Attainment of treatment goals 5 point scale ranging from -2 to 2, higher score representing better outcome
Faces Pain Scale | Post-treatment weeks 4-12-20
  Assessment of pain by a visual 6 point scale ranging from 0 to 10, 0 representing no pain, 10 representing most excruciating pain

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Dursun, MD, Principal Investigator — Kocaeli Universitesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carranza-Del Rio J, Dursun N, Cekmece C, Bonikowski M, Pyrzanowska W, Dabrowski E, Tilton A, Oleszek J, Volteau M, Page S, Shierk A, Delgado MR. Goal Attainment after Treatment with Abobotulinumtoxina and a Tailored Home Therapy Programme in Children with Upper Limb Spasticity: Descriptive, Exploratory Analysis of a Large Randomized, Controlled Study. J Rehabil Med. 2022 Dec 9;54:jrm00349. doi: 10.2340/jrm.v54.2540. PMID 36306168
- [Result] Dursun N, Gokbel T, Akarsu M, Bonikowski M, Pyrzanowska W, Dursun E. Intermittent serial casting for wrist flexion deformity in children with spastic cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2021 Jun;63(6):743-747. doi: 10.1111/dmcn.14765. Epub 2021 Jan 22. PMID 33483965
- [Result] Delgado MR, Tilton A, Carranza-Del Rio J, Dursun N, Bonikowski M, Aydin R, Maciag-Tymecka I, Oleszek J, Dabrowski E, Grandoulier AS, Picaut P; Dysport in PUL study group. Efficacy and safety of abobotulinumtoxinA for upper limb spasticity in children with cerebral palsy: a randomized repeat-treatment study. Dev Med Child Neurol. 2021 May;63(5):592-600. doi: 10.1111/dmcn.14733. Epub 2020 Nov 18. PMID 33206382
- [Result] Dursun N, Gokbel T, Akarsu M, Dursun E. Randomized Controlled Trial on Effectiveness of Intermittent Serial Casting on Spastic Equinus Foot in Children with Cerebral Palsy After Botulinum Toxin-A Treatment. Am J Phys Med Rehabil. 2017 Apr;96(4):221-225. doi: 10.1097/PHM.0000000000000627. PMID 27631386
- [Result] Delgado MR, Tilton A, Russman B, Benavides O, Bonikowski M, Carranza J, Dabrowski E, Dursun N, Gormley M, Jozwiak M, Matthews D, Maciag-Tymecka I, Unlu E, Pham E, Tse A, Picaut P. AbobotulinumtoxinA for Equinus Foot Deformity in Cerebral Palsy: A Randomized Controlled Trial. Pediatrics. 2016 Feb;137(2):e20152830. doi: 10.1542/peds.2015-2830. Epub 2016 Jan 26. PMID 26812925
- [Result] Dursun N, Bonikowski M, Dabrowski E, Matthews D, Gormley M, Tilton A, Carranza J, Grandoulier AS, Picaut P, Delgado MR. Efficacy of Repeat AbobotulinumtoxinA (Dysport(R)) Injections in Improving Gait in Children with Spastic Cerebral Palsy. Dev Neurorehabil. 2020 Aug;23(6):368-374. doi: 10.1080/17518423.2019.1687602. Epub 2019 Nov 6. PMID 31691605
- [Result] Chang MC, Choo YJ, Kwak SG, Nam K, Kim SY, Lee HJ, Kwak S. Effectiveness of Extracorporeal Shockwave Therapy on Controlling Spasticity in Cerebral Palsy Patients: A Meta-Analysis of Timing of Outcome Measurement. Children (Basel). 2023 Feb 9;10(2):332. doi: 10.3390/children10020332. PMID 36832460
- [Result] Mihai EE, Popescu MN, Iliescu AN, Berteanu M. A systematic review on extracorporeal shock wave therapy and botulinum toxin for spasticity treatment: a comparison on efficacy. Eur J Phys Rehabil Med. 2022 Aug;58(4):565-574. doi: 10.23736/S1973-9087.22.07136-2. Epub 2022 Apr 12. PMID 35412036
- [Result] Kwon DR, Kwon DG. Botulinum Toxin a Injection Combined with Radial Extracorporeal Shock Wave Therapy in Children with Spastic Cerebral Palsy: Shear Wave Sonoelastographic Findings in the Medial Gastrocnemius Muscle, Preliminary Study. Children (Basel). 2021 Nov 17;8(11):1059. doi: 10.3390/children8111059. PMID 34828772